CLINICAL TRIAL: NCT02828878
Title: An Open-Label Phase I/II, Pilot, Staggered Four-Cohort Safety and Proof-of-Concept Study of ApoGraft in the Prevention of Acute Graft Versus Host Disease (aGvHD)
Brief Title: Prevention of Acute Graft Versus Host Disease in Patients Undergoing Allogeneic ApoGraft Stem Cell Transplantation
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cellect Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ApoGraft 01
Record Dates: First submitted 2016-07-04; First posted 2016-07-12 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Hematological Malignancies
Keywords: Apoptosis; FAS Ligand; Bone marrow transplantation; GvHD; Stem cells
MeSH Terms: conditions — Hematologic Neoplasms; Autoimmune Lymphoproliferative Syndrome, Type IB

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ApoGraft (Experimental): ApoGraft is a mobilized peripheral blood cell (MPBC) product derived from peripheral blood. There will be 4 cohorts, each differ in the amount of apoptotic mediator Fas Ligand (APO010) to which the graft is exposed during incubation prior to ApoGraft transplant, ranging from 10 ng/ml APO010 in Cohort 1, 25 ng/ml APO010 in Cohort 2, 50 ng/ml APO010 in Cohort 3, and 100 ng/ml APO010 in Cohort 4
  Interventions: Biological: Allogeneic MPBC transplantation from matched related donor

INTERVENTIONS:
Biological: Allogeneic MPBC transplantation from matched related donor

SUMMARY:
Interventional, open label, Phase I/II, Safety and Proof-of-Concept Study, with a follow up period of 180 days after the transplantation of ApoGraft.

DETAILED DESCRIPTION:
ApoGraft product is a mobilized peripheral blood cell product of a matched Related donor, collected via apheresis, which is exposed to the apoptotic mediator Fas Ligand (CD95L) prior to transplantation (Ex Vivo).

The study is designed to address the aspects of engraftment and Prevention of Acute Graft versus Host Disease (aGvHD) rate and/or severity in 12 Patients

STUDY DESIGN:

This is a phase 1/2, open-label, proof-of-concept, staggered 4-cohort clinical study. Each cohort will include 3 patients with hemato-oncology disorders eligible for allogeneic HLA-matched HSCT. Patients in all cohorts will undergo similar study procedures and evaluation. The cohorts will differ from each other in the amount of apoptotic mediator Fas Ligand (APO010) to which the graft is exposed during incubation prior to ApoGraft transplantation and HSCT, ranging from 10 ng/ml APO010 in Cohort 1, 25 ng/ml APO010 in Cohort 2, 50 ng/ml APO010 in Cohort 3 and 100 ng/ml APO010 in Cohort 4. APO010 is washed-out as part of the ApoGraft process and only trace amounts of APO010 are present in the final ApoGraft product

The study consists of a screening phase (subject and donor clinical assessment and screening tests), transplantation of ApoGraft, and a follow-up period of 180 days during and after hospitalization.

The study will progress from one cohort to the next based on an independent data safety monitoring board (DSMB) review and analysis of safety data

ELIGIBILITY:
Recipient/patient main inclusion criteria:

1. Adult male or female subjects, 18-70 years of age.
2. Subjects are eligible for allogeneic HLA-matched related HSCT for any hematological malignancies for which transplantation is appropriate with corresponding related donor. One of the following hemato-oncology disorders diagnosis is required:

   * Acute myelogenous leukemia (AML) and Acute lymphoblastic leukemia (ALL) in 1st or subsequent complete remission (CR)
   * Non-Hodgkin's disease (NHD) in CR by CT or PET/CT
   * Hodgkin's disease (HD) in 1st or subsequent CR by CT or PET/CT
   * Intermediate, High or Very High Risk Myelodysplastic syndrome (MDS) (IPSS-R criteria)
3. The donor and recipient must have full match at the HLA A, B, C, DR and DQ loci.
4. ECOG performance status score 0-1 at time of the screening visit.
5. Subjects must have adequate organ function as defined in the study protocol
6. Signed written informed consent to participate in the study.
7. If female of childbearing potential, agree to use an acceptable method of birth control or be surgically sterile, and have a negative pregnancy test.

Donor main inclusion criteria:

1. Adult male or female subjects, 18-65 years of age.
2. Donor criteria according to standard WMDA criteria for donor selection. 3 Must have full match at the HLA A, B, C, DR and DQ loci with the recipient.

4. Signed written informed consent

Recipient/patient main exclusion criteria:

1. Use of non-myeloabletive conditioning.
2. Uncontrolled infections including sepsis, pneumonia with hypoxemia, persistent bacteremia, or meningitis within two weeks of the screening visit.
3. Current known acute or chronic infection with HBV or HCV.
4. Known human immunodeficiency virus (HIV) infection or AIDS.
5. Subjects with severe or symptomatic restrictive or obstructive lung disease or respiratory failure requiring ventilator support.
6. Subjects with other concurrent severe and/or uncontrolled medical condition, which could compromise participation in the study (i.e. active infection, uncontrolled diabetes, uncontrolled hypertension, congestive cardiac failure, unstable angina, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within six months and chronic liver or renal disease.
7. Any form of substance abuse (including drug or alcohol abuse), psychiatric disorder or any chronic condition susceptible, in the opinion of the investigator, of interfering with the conduct of the study.
8. Organ allograft or previous history of allogeneic stem cell transplantation.
9. Pregnancy or lactation.

Donor main exclusion criteria:

1. HIV, HBV or HCV positive subjects.
2. Pregnant or lactating women.
3. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Overall incidence, frequency and severity of adverse events (AEs) potentially related to the product during the study | 180 days from transplantation

SECONDARY OUTCOMES:
Determination of the optimal dose of FasL concentration that facilitates the biological activity of the ApoGraft process | 180 days from transplantation
Time of neutrophils engraftment determined by number of days for reaching first of 3 consecutive days with ANC ≥ 500/mm3 | 28 days from transplantation
Rate of neutrophils engraftment determined by number of days for reaching first of 3 consecutive days with ANC ≥ 500/mm3 | 28 days from transplantation
Time of platelets engraftment determined by number of days for reaching first of 3 consecutive days with platelets ≥ 20,000/mm3 in the absence of platelet administration during the prior 7 days | 180 days from transplantation
Rate of platelets engraftment determined by number of days for reaching first of 3 consecutive days with platelets ≥ 20,000/mm3 in the absence of platelet administration during the prior 7 days | 180 days from transplantation
Incidence to development of aGvHD | 180 days from transplantation
Time to development of aGvHD | 180 days from transplantation
Non-relapse mortality | 180 days from transplantation
Proportion of patients with disease relapse | 180 days from transplantation
Proportion of patients with progression free and overall survival | 180 days from transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Tsila Zuckerman, MD, Principal Investigator — Rambam Hospital, Haifa, Israel
Locations (2):
- Israel (2):
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center, Ein Kerem, Jerusalem, Jerusalem

IPD SHARING:
Plan to Share IPD: No